CLINICAL TRIAL: NCT05062382
Title: Complementary Feeding Project in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Global Alliance for Improved Nutrition (Other)
Responsible Party: Principal Investigator, Edward Frongillo, Jr., Principal Investigator, University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 102
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Egg Consumption

STUDY DESIGN:
Intervention Model Description: Cross-sectional pre- post-evaluation of intervention and comparison group
Who Masked: Outcomes Assessor
Masking Description: Data collectors were masked to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complementary feeding program (Experimental): Promotion of eggs.
  Interventions: Behavioral: Complementary feeding intervention
- Comparison (No Intervention): Comparison arm with no program

INTERVENTIONS:
Behavioral: Complementary feeding intervention — The study promoted eggs.
  GAIN provided training to egg farmers to increase their egg production and marketing, helped increase mother's access to eggs by making them more available in local kiosks and getting retailers to display promotional messages around eggs, conducted sensitization workshops with retailers to increase egg purchases, and employed a demand creation campaign.
  Arms: Complementary feeding program

SUMMARY:
The Global Alliance for Improved Nutrition (GAIN), a Swiss-based foundation, implemented a complementary feeding project to improve dietary quality among children 6-59 months of age living in Ethiopia by improving demand and access to eggs. Using a quasi-experimental design and two separate cross-sectional surveys at baseline and end-line, the evaluation seeks to determine the effects of the program on egg consumption, availability of eggs, caregivers' behaviours toward eggs, and caregivers' willingness to pay for eggs.

DETAILED DESCRIPTION:
The Global Alliance for Improved Nutrition (GAIN), a Swiss-based foundation, implemented a complementary feeding project to improve dietary quality among children 6-59 months of age living in Ethiopia by improving demand and access to eggs. The complementary feeding project aimed to boost children's consumption of eggs. The intervention incorporated demand creation campaigns and supported selected delivery channels and producers who provided eggs to communities. GAIN's demand creation strategy was designed to complement the Ethiopian government's effort to use social and behavior change communication to encourage consumption of nutritious complementary foods. This campaign was implemented through the existing health extension system.

Areas included in the intervention arm received direct support for egg producers and suppliers and an egg demand creation campaign. Supply-side interventions included training for farmers, identification of distribution channels, mapping of retailers, and creation of linkages between egg producers and egg suppliers. Egg demand-creation activities were executed through above-the-line (ATL) and below-the-line (BTL) campaigns. The ATL campaigns included radio messages, bajaja branding, billboard mounting, and digital promotion. The BTL campaigns include market activation, road shows, sensitization workshops for key community groups, door-to-door promotion, and mobile promotion in collaboration with creative agencies and health extension workers. Both sets of activities focused on creating awareness around eggs as a daily nutritious food option for children.

Originally, the study intended to also increase availability of, and demand for, commercially-available complementary foods (i.e., Cerifam and Fafa), however, these components of the intervention were not delivered. Therefore, we have removed these components from the description and removed the outcomes that corresponded with these components of the intervention.

Using a quasi-experimental design and two separate cross-sectional surveys at baseline and end-line, the evaluation seeks to determine the effects of the program on egg consumption, availability of eggs, caregivers' behaviours toward eggs, and caregivers' willingness to pay for eggs.

ELIGIBILITY:
Inclusion Criteria:

* Living in the project areas
* Caregiver 18 years old or above

Exclusion Criteria:

* households without children between the ages of 6-59 months

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1132 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in the number of eggs consumed from baseline to end-line | From baseline to 22 months
  Change in the average number of eggs consumed in the past 7 days by children 6 to 59 months of age from baseline to end-line in the two study arms
Change in the consumption of eggs from baseline to end-line | From baseline to 22 months
  Change in the proportion of children 6-59 months of age consuming eggs in the last 7 days and in the last 24 hours from baseline to end-line in the two study arms

SECONDARY OUTCOMES:
Change in household egg production from baseline to end-line | From baseline to 22 months
  Change in the proportion of households producing eggs from baseline to end-line in the two study arms
Change in egg purchasing from baseline to end-line | From baseline to 22 months
  Change in the proportion of households that purchased egg in the last month from baseline to end-line in the two study arms
Change in caregivers' (of children 6-59 months) behavioral determinants in the context of feeding eggs to children from baseline to end-line | From baseline to 22 months
  Change in the mean factor score created from Likert scales of attitudes (attitudes scale, higher score reflects better attitudes towards eggs), norms (norms scale, higher score reflects better norms towards eggs), self-efficacy (self-efficacy scale, higher score reflects better self-efficacy), and intention towards eggs (intent to feed eggs to child, higher score reflects more intent to feed eggs) from baseline to end-line between the two study arms; change will be examined for a meta factor score combining all scales and each scale separately. Values of factor scores are unbounded and can be positive or negative.
Change in caregivers' willingness to pay for eggs from baseline to end-line | From baseline to 22 months
  Change in willingness to pay for eggs, using for example the change in mean maximum price that caregivers would be willing to pay for eggs from baseline to endline between the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Frongillo, PhD, Principal Investigator — University of South Carolina
Locations (1):
- Deep Dive Research and Consulting PLC, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Reports will be made available. We will provide information on how to make the request to have access to the partial or complete anonymized dataset.
Supporting Information: CSR